CLINICAL TRIAL: NCT04605627
Title: The Role of Gut Leakage Markers and Microbiota Signature in Coronary Artery Disease.
Acronym: GUT-ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Geir Øystein Andersen, MD, PhD, Senior Cardiologist, Oslo University Hospital
Other Study IDs: Oslo University Hospital
Record Dates: First submitted 2020-09-30; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease; Intestinal Disease
Keywords: Gut leakage; Microbiota; Coronary artery disease; STEMI; NSTEMI; Chronic coronary syndrome
MeSH Terms: conditions — Coronary Artery Disease; Intestinal Diseases; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Peripheral blood mononuclear cells (PBMC), feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic coronary syndrome: 50 patients with chronic coronary disease
- Non ST segment-elevation myocardial infarction: 75 patients with non ST-elevation myocardial infarction
- ST-elevation myocardial infarction: 75 patients with ST segment-elevation myocardial infarction

SUMMARY:
Define a signature of gut microbiota composition and related metabolites in patients with ST-elevation myocardial infarction, non ST-elevation myocardial infarction and chronic coronary disease (CAD).

DETAILED DESCRIPTION:
A total of 200 patients, allocated to 50 patients with chronic coronary syndrome, 75 patients with non-ST elevation myocardial infarction and 75 patients with ST- elevation myocardial infarction will be included. Clinical information, blood samples and fecal samples will be collected. Fecal and blood samples will be collected once in patients With chronic disease and in patients with acute coronary syndrome; in the acute phase and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease verified by coronary angiography

Exclusion Criteria:

* Current infection requiring intravenous antibiotics
* Inflammatory bowel disease
* Renal failure with creatinine > 200µmol/L
* Hepatic impairment
* Pregnancy
* Previous bariatric surgery
* Colostomy
* Active malignant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20-75 years with coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota alpha diversity in myocardial infarction measured as Chao1 Index. | Within 7 days from inclusion.
  fecal-sample. 16srRNA (Miseq) will be used for sequencing.
Microbiota alpha diversity in myocardial infarction measured as Chao1 Index | At 3 months follow-up.
  fecal-sample. 16srRNA (Miseq) will be used for sequencing.
Lipopolysaccharide binding protein (LBP) in myocardial infarction | At inclusion
  Blood sample. Analyses will be performed with ELISA.
Lipopolysaccharide binding protein (LBP) in myocardial infarction | Change from inclusion to 3 months follow-up.
  Blood sample. Analyses will be performed with ELISA.
Soluble cluster of difference-14 in myocardial infarction | At inclusion
  Blood sample. Analyses will be performed with ELISA.
Soluble cluster of difference-14 in myocardial infarction | Change from inclusion to 3 months follow-up.
  Blood sample. Analyses will be performed with ELISA.
Intestinal fatty acid binding protein-1 in myocardial infarction | At inclusion
  Blood sample. Analyses will be performed with ELISA.
Intestinal fatty acid binding protein-1 in myocardial infarction | Change from inclusion to 3 months follow-up.
  Blood sample. Analyses will be performed with ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Trøseid, Md Ass.prof, Principal Investigator — Oslo University Hospital
Locations (1):
- Department of Cardiology, Oslo University Hospital Ullevål, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, informed consent form (in Norwegian) and clinical study report will be shared by request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data become available 01.06.2022, and will be available until 01.06.2023.
Access Criteria: Requests by email will be answered.